CLINICAL TRIAL: NCT03045159
Title: Supporting Military Families With Young Children Throughout the Deployment Lifecycle
Brief Title: Strong Families Strong Forces: Supporting Active Duty Families With Very Young Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston University (Other)
Collaborators: The University of Texas Health Science Center at San Antonio (Other); RAND (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: W81XWH-14-2-0123
Record Dates: First submitted 2016-03-31; First posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2016-03

CONDITIONS: Deployment
Keywords: deployment cycle; military family; prevention; stress; military child; parenting; coparenting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: outcomes assessor blinded to study condition
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Strong Families (Experimental): parenting program
  Interventions: Behavioral: Strong Families Strong Forces
- Strong Parents (Active Comparator): self-care program
  Interventions: Behavioral: Strong Parents

INTERVENTIONS:
Behavioral: Strong Families Strong Forces — Parenting program
  Arms: Strong Families
Behavioral: Strong Parents — self-care program
  Arms: Strong Parents

SUMMARY:
The purpose of this research is to evaluate the efficacy of the Strong Families Strong Forces Parenting Program compared to a parental self-care (Strong Parents) condition in a sample of 150 Active Duty Families with children ages birth to 5 years.

DETAILED DESCRIPTION:
The overall aim of this research is to adapt and evaluate the efficacy of a parenting program compared to a parental self-care program for Active Duty families. A sample of 150 Active Duty families with young children who have a parent scheduled to deploy in the next six months will be recruited to participate. Families will be assigned either to receive the Strong Families Strong Forces Parenting Program, designed to reduce the impact of deployment separation on parenting stress and co-parenting, or to the Strong Parents Self-Care program, designed to support parents to focus on the importance of self-care throughout the deployment cycle. Investigators will compare the two groups on parenting stress, quality of parent-child relationships, parenting/co-parenting, and family and child well-being.

ELIGIBILITY:
Inclusion Criteria:

* Cohabitating couple with at least one child age birth to 5 years old in which one parent is active duty and is scheduled to deploy within the next 6 months
* Anticipated deployment time must be at least six months and excludes separations due to the Service Member attending a school
* Anticipate that non-deploying parent will remain in the area during the deployment
* Both parents are willing to consent to study participation
* DEERS -eligible
* 18 years or older
* English-speaking
* The parent remaining at home to care for the children anticipates remaining within 30 miles of Fort Hood to be seen in home, otherwise will need to be seen in office
* Anticipate that both parents will remain in the area for at least three months after redeployment to complete intervention and follow-up assessment

Exclusion Criteria:

* Any family member with a significant medical or psychiatric condition requiring a higher level of care than can be provided by the study/comparison protocols
* Active psychosis or mania

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Parenting Stress Index (PSI) | Change from baseline to 24 months
  Assesses parenting stress in three domains: parental distress, parent-child dysfunctional interaction, and difficult child.

SECONDARY OUTCOMES:
Coparenting Scale | Change from baseline to 24 months
  Assesses parents' perception of their own coparenting behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen DeVoe, Ph. D. LICSW, Principal Investigator — Boston University
Locations (1):
- STRONG STAR Research Consortium, Fort Hood, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided